CLINICAL TRIAL: NCT07381803
Title: The Impact of Fexofenadine Hydrochloride on the Prognosis of Patients Post-Acute Myocardial Infarction: A Randomized Clinical Trial (FEND Ⅱ)
Brief Title: The Impact of Fexofenadine Hydrochloride on the Prognosis of Patients Post-Acute Myocardial Infarction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YAN2025-1734
Record Dates: First submitted 2026-01-05; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-01

CONDITIONS: Zhejiang University
Keywords: myocardial infarction; cardiac fibrosis; cardiac MRI
MeSH Terms: conditions — Myocardial Infarction | interventions — fexofenadine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fexofenadine (Experimental): 60mg, BID
  Interventions: Drug: Fexofenadine 60 Mg Oral Tablet

INTERVENTIONS:
Drug: Fexofenadine 60 Mg Oral Tablet — Fexofenadine, 60mg BID oral
  Arms: Fexofenadine
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The goal of this study is o evaluate the prognostic effect of fexofenadine hydrochloride in patients with myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Able to verbally confirm understanding of the trial risks, benefits, and treatment options of fexofenadine hydrochloride therapy. He/she or his/her legal representative must provide written informed consent prior to participating in the clinical trial.
* Acute ST-segment elevation myocardial infarction (STEMI) occurring within 7 days, with diagnostic criteria including:

  i) Typical clinical symptoms: such as severe crushing pain in the retrosternal or precordial area, usually lasting more than 10-20 minutes, which may radiate to the left upper arm, jaw, neck, back, or shoulders, etc.; ii) Elevated serum cardiac troponin (cTn): at least one measurement above the upper limit of normal (99th percentile of the reference upper limit); iii) ST-segment elevation: new ST-segment elevation at the J point in 2 adjacent leads.
* Echocardiography indicating segmental wall motion abnormalities.

Exclusion Criteria:

* Need for long-term use of fexofenadine hydrochloride or other H1 receptor inhibitors.
* Previous coronary artery bypass grafting (CABG) surgery.
* History of severe renal failure with estimated glomerular filtration rate (eGFR) < 30 ml/min.
* History of severe liver dysfunction.
* History of concurrent severe infection, hepatobiliary obstruction, or malignant tumor.
* Expected life expectancy of less than 2 years due to non-cardiac diseases.
* Currently receiving immunosuppressive therapy.
* Pregnant, potentially pregnant, or lactating women.
* Contraindication to the study drug or examinations.
* Failure to provide written informed consent.
* Presence of mechanical complications (ventricular septal defect, papillary muscle dysfunction, acute mitral regurgitation), refractory cardiogenic shock unresponsive to vasopressors, acute left heart failure or pulmonary edema, or malignant arrhythmias uncontrolled by antiarrhythmic drugs at enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2804 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | 24 months
  MACCE within 24 months after randomization, including all-cause death, recurrent myocardial infarction, stroke, hospitalization for heart failure, outpatient or emergency visits due to worsening heart failure, and repeat revascularization driven by angina pectoris.

SECONDARY OUTCOMES:
All-cause death | 24 months, 60 months after myocardial infarction
  All-cause death between 2 groups
Recurrent myocardial infarction | 24 and 60 months after myocardial infarction
  Recurrent myocardial infarction between 2 groups
Stroke | 24 and 60 months after myocardial infarction
  Stroke incidence between 2 groups
Hospitalization for heart failure | 24 and 60 months after myocardial infarction
  The incidence of Hospitalization for heart failure between 2 groups
Repeat revascularization driven by angina pectoris | 24 and 60 months after myocardial infarction
  Repeat revascularization driven by angina pectoris between 2 groups
Left ventricular ejection fraction (LVEF%) | 24 months after myocardial infarction
  Comparison of the difference in left ventricular ejection fraction (LVEF%) measured by echocardiography between the two groups at 24 months after randomization compared to baseline.
Left ventricular end-systolic diameter (LVIDs) | 24 months after myocardial infarction
  Comparison of the difference in left ventricular end-systolic diameter (LVIDs) measured by echocardiography between the two groups at 24 months after randomization compared to baseline.
Left ventricular end-diastolic diameter (LVIDd) | 24 months after myocardial infarction
  Comparison of the difference in left ventricular end-diastolic diameter (LVIDd) measured by echocardiography between the two groups at 24 months after randomization compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

DOCUMENTS (1):
  • Study Protocol (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT07381803/Prot_000.pdf